CLINICAL TRIAL: NCT04667299
Title: Bismuth-Metronidazole Triple Versus Quadruple Therapy for Helicobacter Pylori First-line Treatment: A Randomized Controlled Trial
Brief Title: Bismuth-Metronidazole Triple Therapy for H. Pylori First-line Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2020-261
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Rabeprazole; Metronidazole; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMT group (Experimental): Rabeprazole 20 mg bid, bismuth potassium citrate 0.6 g bid and metronidazole 0.4 g qid for 14 days
  Interventions: Drug: Rabeprazole; Drug: Bismuth potassium citrate; Drug: Metronidazole
- BMQ group (Active Comparator): Rabeprazole 20 mg bid, bismuth potassium citrate 0.6 g bid, metronidazole 0.4 g qid and amoxicillin 1 g bid for 14 days
  Interventions: Drug: Rabeprazole; Drug: Bismuth potassium citrate; Drug: Metronidazole; Drug: Amoxicillin

INTERVENTIONS:
Drug: Rabeprazole — 20mg bid
Drug: Bismuth potassium citrate — 0.6g bid
Drug: Metronidazole — 0.4g qid
Drug: Amoxicillin — 1g bid
  Arms: BMQ group

SUMMARY:
This randomized controlled clinical trial will compare the eradication efficacy of bismuth-metronidazole triple therapy (PPI+bismuth+ metronidazole) with that of bismuth-metronidazole quadruple therapy (PPI+bismuth+ metronidazole+ amoxicillin) for Helicobacter pylori first-line treatment. The completion of this trial will expand new therapy for the treatment of Helicobacter pylori, which can not only ensure clinical efficacy, but also reduce the use of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Participate in the trial voluntarily, fully understand the trial, and sign the informed consent form (ICF).
* 18-75 years old on the day of signing the ICF.
* Helicobacter pylori infection confirmed by 13C-urea breath test or rapid urease test.
* Have not received Helicobacter pylori eradication treatment before.

Exclusion Criteria:

* Have received Hp eradication treatment.
* Patients with severe heart, lung, kidney, liver, blood, nerve, endocrine, and psychiatric diseases.
* Subjects or guardians refused to participate in the trial.
* Alcohol and/or drugs Abuse (addiction or dependence) or poor compliance with doctor's judgment.
* Have taken antibiotics, bismuth, PPI or Chinese traditional medicine 4 weeks before treatment.
* Pregnant or lactating women.
* Active peptic ulcer.
* allergic to drugs used in the trial.
* any other circumstances that are not suitable for recruitment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori | At least 4 weeks after completion of therapy
  Eradication of Helicobacter pylori was defined as negative result of urea breath test (<4‰ cut-off value).

SECONDARY OUTCOMES:
Eradication rate of Helicobacter pylori metronidazole-resistant strains | At least 4 weeks after completion of therapy
  Eradication of Helicobacter pylori was defined as negative result of urea breath test (<4‰ cut-off value). The strains with minimal inhibitory concentration (MIC) value of metronidazole >8 μg/ml were defined as resistant strains.
Eradication rate of Helicobacter pylori metronidazole-susceptible strains | At least 4 weeks after completion of therapy
  Eradication of Helicobacter pylori was defined as negative result of urea breath test (<4‰ cut-off value). The strains with metronidazole MIC value <=8 μg/ml were defined as susceptible strains.

OTHER OUTCOMES:
Adherence rate | At least 1 weeks after completion of therapy
  Adherence was defined as poor when subjects took less than 80% of the total medication.
Frequency of adverse events | At least 1 weeks after completion of therapy
  Any possible adverse events during the 14-day treatment period were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Taotao Liu, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be available from the principal investigator Taotao Liu at liu.taotao@zs-hospital.sh.cn, beginning 6 months and ending 5 years after the trial results were published. The study protocol and statistical analysis plan are available online from https://clinicaltrials.gov/. All proposals requesting data access will need to specify how it is planned to use the data, and all proposals will need approval of all investigators before data release.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 5 years after the trial results were published.
Access Criteria: All proposals requesting data access will need to specify how it is planned to use the data, and all proposals will need approval of all investigators before data release.
URL: http://clinicaltrials.gov/